CLINICAL TRIAL: NCT02427555
Title: Effects of Barley Based Food Products on Metabolism and Gut Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AFC-Y8-2015
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Subjects

ARMS (2):
- Barley kernel bread (Experimental)
  Interventions: Other: Barley kernel bread
- Whit wheat flour bread (Sham Comparator)
  Interventions: Other: white wheat bread

INTERVENTIONS:
Other: Barley kernel bread — 3 days intervention with barley kernel bread
  Arms: Barley kernel bread
Other: white wheat bread — 3 days intervention with white wheat bread
  Arms: Whit wheat flour bread

SUMMARY:
The main objective is to investigate gut microflora composition in relation to cardiometabolic risk markers, and to investigate the effects of 3 days intervention with a barley kernel based product on these variables.

DETAILED DESCRIPTION:
100 subjects were invited to deliver faecal samples. From this cohort 40 subjects were chosen based on their gut microflora composition to participate in the Barley intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women between 50-79 years and
* BMI between 19-28.

Exclusion Criteria:

* fasting blood glucose concentrations > 6,1 mmol/L,
* known metabolic disorders or gastrointestinal diseases or other disorders that can interfere with the results of the study.
* furthermore, the subjects should be non-smokers and
* consume a normal (non-vegetarian) diet as is recommended by the Nordic dietary guidelines.
* antibiotics or probiotics should not have been taken during four weeks prior to faeces donation.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in glucose regulation | Changes in fasting and postprandial blood glucose concentrations after 3 days intervention with a barley based bread in comparison to 3 days intervention with a white wheat based bread
  blood glucose concentrations are measured fasting and postprandially a standardised breakfast after interventions with barley based bread and white wheat bread, respectively
Changes in colonic microbiota composition after intervention with barley | Changes in colonic microbiota composition after 3 days intervention with a barley based bread in comparison to 3 days intervention with a white wheat based bread
  Gut microbiota composition are characterised after interventions with barley based bread and white wheat bread, respectively
nucleotide polymorphisms (SNP in TCF7L2) | at baseline
  investigate nucleotide polymorphisms that associate with cardiometabolic traits, in particular the SNP in TCF7L2

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Food for Health Science Centre, Medicon Village, Lund University
Locations (1):
- Food for Health Science Centre, Medicon Village, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Sandberg J, Kovatcheva-Datchary P, Bjorck I, Backhed F, Nilsson A. Abundance of gut Prevotella at baseline and metabolic response to barley prebiotics. Eur J Nutr. 2019 Sep;58(6):2365-2376. doi: 10.1007/s00394-018-1788-9. Epub 2018 Jul 25. PMID 30046942